CLINICAL TRIAL: NCT00317356
Title: A Dose-finding Study of OPC-6535 in Patients With Active Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Efficacy was not cleared at US study
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 197-05-002; JapicCTI-060216
Record Dates: First submitted 2006-04-21; First posted 2006-04-24 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Colitis, Ulcerative
Keywords: OPC-6535; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — tetomilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: OPC-6535(Tetomilast)

SUMMARY:
The purpose of this study is to examine the safety and efficacy of OPC-6535 (tetomilast) and to determine its optimal dose by once-daily oral administration at 0, 12.5, 25, or 50 mg for 8 weeks in combination with a fixed oral dose of 5-aminosalicylic acid (5-ASA) in patients with active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active ulcerative colitis
* Patients who have been receiving an oral 5-ASA formulation at a fixed regimen and at a fixed dose
* Either inpatient or outpatient

Exclusion Criteria:

* Patients who have a history of intestinal resection (other than appendiceal resection)
* Patients who have a complication of malignant tumor
* Female patients who are pregnant, lactating, or possibly pregnant, or who wish to become pregnant during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Division of New Product Evaluation and Development
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Touhoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-6535 12.5 mg: 12.5 mg OPC-6535 orally administered once daily in the morning for 8 weeks.
- OPC-6535 25 mg: 25 mg OPC-6535 orally administered once daily in the morning for 8 weeks.
- OPC-6535 50 mg: 25 mg OPC-6535 orally administered for the first week and then the dose was increased to 50 mg for the following 7 weeks.
- Placebo: 0 mg OPC-6535 orally administered once daily in the morning for 8 weeks.
Period: Overall Study
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Started | 11 | 11 | 10 | 11
Completed | 10 | 9 | 9 | 8
Not Completed | 1 | 2 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 10 | 11 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 1 | 1
  Between 18 and 65 years | 11 | 11 | 10 | 10 | 42
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 3 | 5 | 19
  Male | 6 | 5 | 7 | 6 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 11 | 11 | 10 | 11 | 43
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 11 | 11 | 10 | 11 | 43

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement Rate (Number of Subjects Showing Clinical Improvement/Number of Subjects Evaluated x 100) After 8 Weeks of Study Drug Administration
Description: Definition of clinical improvement: Disease Activity Index (DAI) subscore for rectal bleeding improved to 0 or 1 and DAI subscore for mucosal appearance improved by at least 1 point from baseline
Time Frame: Weeks 4 and 8
Population: Efficacy was evaluated in the subjects who took at least one dose of the study drug and provided postdosing data concerning the efficacy endpoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 10 | 11
percentage of participants | 27.3 [6.0 to 61.0] | 30.0 [6.7 to 65.2] | 50.0 [18.7 to 81.3] | 9.1 [0.2 to 41.3]

2. Secondary Outcome: Remission Rate (Number of Subjects Showing Remission/Number of Subjects Evaluated x 100) After 4 and 8 Weeks of Study Drug Administration
Description: Definition of remission: DAI subscores for both rectal bleeding and mucosal appearance improved to 0
Time Frame: Weeks 4 and 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 10 | 11
percentage of participants
  Week 4 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 36.9] | 9.1 [0.2 to 41.3]
  Week 8 | 0.0 [0.0 to 28.5] | 9.1 [0.2 to 41.3] | 10.0 [0.3 to 44.5] | 9.1 [0.2 to 41.3]

3. Secondary Outcome: Mean Change From the Baseline in Total DAI Score After 4 and 8 Weeks of Study Drug Administration
Description: DAI measures disease activity through assessment of 4 items/subscales: stool frequency, rectal bleeding, mucosal appearance at endoscopy, and physician's rating of disease activity. Each item of the score is assessed on a 4-point scale from 0 to 3; the total score ranges from 0 to 12 with a higher score representing greater severity. A negative change in mean score indicates improvement.
Time Frame: Baseline, Weeks 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 10 | 11
score on a scale
  Week 4: number analyzed (Participants) | 4 | 3 | 1 | 3
  Week 4 | -2.5 (2.4) | -1.0 (3.0) | -5.0 | -2.3 (4.2)
  Week 8: number analyzed (Participants) | 10 | 10 | 9 | 9
  Week 8 | -2.6 (2.2) | -1.9 (3.4) | -3.8 (2.2) | -1.4 (2.3)

4. Secondary Outcome: Mean Change From the Baseline in DAI Subscores After 4 and 8 Weeks of Study Drug Administration
Description: DAI measures disease activity through assessment of 4 items/subscales: stool frequency, rectal bleeding, mucosal appearance at endoscopy, and physician's rating of disease activity. Each item of the score is assessed on a 4-point scale from 0 to 3 with a higher score representing greater severity. A negative change in mean score indicates improvement.
Time Frame: Baseline, Weeks 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 10 | 11
score on a scale
  Rectal bleeding at Week 4 | -0.6 (0.8) | -1.0 (1.1) | -0.9 (0.7) | -0.4 (0.7)
  Rectal bleeding at Week 8 | -0.7 (0.9) | -0.9 (1.1) | -1.1 (0.9) | -0.5 (0.7)
  Mucosal appearance at Week 4: number analyzed (Participants) | 4 | 3 | 1 | 3
  Mucosal appearance at Week 4 | -0.5 (0.6) | -0.3 (0.6) | -1.0 | -0.7 (1.2)
  Mucosal appearance at Week 8: number analyzed (Participants) | 10 | 10 | 9 | 9
  Mucosal appearance at Week 8 | -0.7 (0.7) | -0.5 (0.7) | -0.8 (0.7) | -0.3 (0.7)
  Stool frequency at Week 4 | -0.4 (1.0) | -0.8 (1.2) | -0.8 (0.8) | -0.4 (0.7)
  Stool frequency at Week 8 | -0.5 (1.1) | -0.3 (1.3) | -0.6 (0.7) | -0.4 (0.8)
  Physician's rating of disease activity at Week 4 | -0.5 (0.7) | -0.7 (1.0) | -0.9 (0.7) | -0.4 (0.7)
  Physician's rating of disease activity at Week 8 | -0.5 (0.5) | -0.5 (0.9) | -1.0 (0.7) | -0.2 (0.8)

5. Secondary Outcome: Mean Change From the Baseline in Total Clinical Activity Index (CAI) Score After 2, 4, and 8 Weeks of Study Drug Administration
Description: CAI composed of 7 variables: number of stool weekly, blood in stools (weekly average), investigator's global assessment of symptomatic state, abdominal pain/cramps, temperature due to colitis, extraintestinal manifestations, and laboratory findings. The scores ranging from 0 to 29 points (higher scores meaning more severe disease).
Time Frame: Baseline, Weeks 2, 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 10 | 11
score on a scale
  Week 2: number analyzed (Participants) | 11 | 10 | 10 | 11
  Week 2 | -1.2 (3.1) | -2.4 (3.7) | -1.8 (1.5) | -1.0 (1.8)
  Week 4: number analyzed (Participants) | 11 | 10 | 10 | 11
  Week 4 | -1.4 (2.3) | -2.6 (4.1) | -2.9 (2.3) | -1.1 (2.3)
  Week 8: number analyzed (Participants) | 11 | 10 | 10 | 11
  Week 8 | -1.9 (2.2) | -2.6 (3.9) | -3.4 (2.5) | -1.0 (2.5)

6. Secondary Outcome: Mean Change From the Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Score After 8 Weeks of Study Drug Administration
Description: The IBDQ has been frequently adopted in Japanese and overseas clinical assessments as a scale for evaluating the quality of life (QOL) of subjects with inflammatory bowel disease. The IBDQ score was calculated as the sum of the responses (each ranging from 1 to 7) to all 32 questions that address symptoms as a result of Crohn's disease: bowel symptoms, systemic symptoms, emotional function, and social function. Total IBDQ score ranges from 32 to 224 with a higher score indicating a better QOL.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 10 | 11
score on a scale | 22.5 (26.5) | 7.1 (44.3) | 16.0 (40.2) | 9.3 (32.9)

7. Secondary Outcome: Mean Change From the Baseline in IBDQ Subscale Scores After 8 Weeks of Study Drug Administration
Description: The IBDQ has been frequently adopted in Japanese and overseas clinical assessments as a scale for evaluating the quality of life (QOL) of subjects with inflammatory bowel disease. The IBDQ includes 32 items, which are divided into four subscales: bowel symptoms, systemic symptoms, emotional function and social function, and each item is scored on a 7-point scale, ranging from 1 (worst) to 7 (best). Total IBDQ score ranges from 32 to 224 with a higher score indicating a better QOL.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 10 | 11
score on a scale
  Bowel symptoms at Week 8 | 9.3 (12.2) | 4.5 (18.6) | 5.8 (13.4) | 4.5 (11.0)
  Systemic symptoms at Week 8 | 4.5 (5.6) | -1.1 (8.5) | 2.2 (7.0) | 0.0 (5.9)
  Emotional function at Week 8 | 5.5 (8.6) | 1.2 (12.9) | 5.8 (15.0) | 4.0 (10.9)
  Social function at Week 8 | 3.2 (6.1) | 2.5 (8.7) | 2.2 (7.2) | 0.7 (8.8)

8. Secondary Outcome: Clinical Improvement Rate After 4 Weeks of Study Drug Administration
Description: Definition of clinical improvement: DAI subscore for rectal bleeding improved to 0 or 1 and DAI subscore for mucosal appearance improved by at least 1 point from baseline
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 10 | 11
percentage of participants | 12.5 [0.3 to 52.7] | 20.0 [0.5 to 71.6] | 14.3 [0.4 to 57.9] | 10.0 [0.3 to 44.5]

ADVERSE EVENTS:
Time Frame: Treatment period (8 weeks)
Description: Safety was evaluated in the subjects who took at least one dose of the study drug and provided postdosing data concerning the safety endpoints.
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 2/11 | 2/10 | 1/11
Other Adverse Events (participants affected / at risk) | 6/11 | 7/11 | 7/10 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-6535 12.5 mg (N=11) | OPC-6535 25 mg (N=11) | OPC-6535 50 mg (N=10) | Placebo (N=11)
Colitis ulcerative (Gastrointestinal disorders) | 0 | 2 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-6535 12.5 mg (N=11) | OPC-6535 25 mg (N=11) | OPC-6535 50 mg (N=10) | Placebo (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Faeces hard (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 4 | 2 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Feeling abnormal (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 3
Blood potassium decreased (Investigations) | 0 | 1 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 1 | 3 | 1 | 0
Protein urine present (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 3 | 3 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No